CLINICAL TRIAL: NCT01089881
Title: The Effectiveness of 18F-fluorocholine PET in Detecting, Staging and Following-up Prostate Cancer
Brief Title: The Effectiveness of 18F-fluorocholine Positron Emission Tomography (PET) in Detecting, Staging and Following-up Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Hong-Jeng Yu, National Taiwan University Hospital
Other Study IDs: 200706006M
Record Dates: First submitted 2010-03-17; First posted 2010-03-19 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; 18F-fluorocholine; PET; recurrence; metastases
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: patients with BPH
- Group 2: patients with newly diagnosed prostate cancer
- Group 3: patients who have received curative treatment for prostate cancer and are suspicious of recurrence/metastases because of a persistent increase in their serum PSA.

SUMMARY:
Choline is one of the components of phosphatidylcholine, an essential element of phospholipids in the cell membrane. Some malignant cells show their ability to actively incorporate choline to produce phosphocholine and phosphatidylcholine to facilitate tumor cell duplication. The efficacy of 18F-fluorocholine (18F-FCH) for localizing primary or metastatic prostate cancer has been recently reported in limited studies. This study will be conducted to delineate the effectiveness of 18F-FCH PET in (1) differentiating benign prostate hypertrophy (BPH) from prostate cancer, (2) staging prostate cancer, (3) following-up patients with prostate cancer after initial curative therapy.

DETAILED DESCRIPTION:
Background:

Prostate cancer is a leading cause of cancer death for male in Taiwan. Although 18F-FDG PET has been shown to be an effective tool in diagnosing many malignancies, previous studies have shown that 18F-FDG is not a suitable PET tracer for detecting prostate cancer. Choline is one of the components of phosphatidylcholine, an essential element of phospholipids in the cell membrane. Some malignant cells show their ability to actively incorporate choline to produce phosphocholine and phosphatidylcholine to facilitate tumor cell duplication. The efficacy of 18F-fluorocholine (18F-FCH) for localizing primary or metastatic prostate cancer has been recently reported in limited studies.

Purpose:

This study will be conducted to delineate the effectiveness of 18F-FCH PET in (1) differentiating benign prostate hypertrophy (BPH) from prostate cancer, (2) staging prostate cancer, (3) following-up patients with prostate cancer after initial curative therapy.

Patients and Methods:

This study will include

1. Group 1: 50 patients with BPH
2. Group 2: 50 patients with newly diagnosed prostate cancer and
3. Group 3: 50 patients who have received curative treatment for prostate cancer and are suspicious of recurrence/metastases because of a persistent increase in their serum PSA.

18F-FCH whole-body PET will be performed for each patient

Expected Results:

To evaluate the effectiveness of 18F-FCH in the diagnosis, staging and follow-up of prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

Group 1: 50 patients with BPH

1. Age above 35 years old
2. Histologically confirmed BPH
3. Informed consent signed

Group 2: 50 patients with newly diagnosed prostate cancer and

1. Age above 35 years old
2. Histologically confirmed prostate cancer
3. Informed consent signed

Group 3: 50 patients who have

1. Age above 35 years old
2. Histologically confirmed prostate cancer and had received curative treatment for prostate cancer
3. suspicious of recurrence/metastases because of a persistent increase in their serum PSA
4. Informed consent signed

Exclusion Criteria:

* Patients with other known malignancies will be excluded.

Ages: 35 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Group 1: 50 patients with BPH
  2. Group 2: 50 patients with newly diagnosed prostate cancer and
  3. Group 3: 50 patients who have received curative treatment for prostate cancer and are suspicious of recurrence/metastases because of a persistent increase in their serum PSA.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hong Jeng, M.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan